CLINICAL TRIAL: NCT02394002
Title: The Effect of Burst-suppression-pattern in EEG on Generating Somatosensory Evoked Potentials
Brief Title: SEP Changes During Deep Anesthesia
Acronym: SEPinBSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andrea Szelenyi (Other)
Collaborators: Department of Anaesthesiology, Heinrich Heine University (Unknown); Department of Anesthesiology, Helios Klinikukm Wuppertal (Unknown)
Responsible Party: Sponsor-Investigator, Andrea Szelenyi, Prof. Dr. med. Andrea Szelényi, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013071151
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Somatosensory Evoked Potentials, and Electroencephalography
Keywords: EEG, burst-suppression, N20, SEP, median nerve, facilitation
MeSH Terms: interventions — Propofol

ARMS (3):
- Brain surgery (Experimental): Somatosensory evoked potentials in relation to anasthesia (Propofol bolus) induced burst and suppression periods in electroencephalography
  Interventions: Drug: Propofol
- Spine surgery (Experimental): Somatosensory evoked potentials in relation to anasthesia (Propofol bolus) induced burst and suppression periods in electroencephalography
  Interventions: Drug: Propofol
- General surgery (Active Comparator): Somatosensory evoked potentials in relation to anasthesia (Propofol bolus) induced burst and suppression periods in electroencephalography
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol

SUMMARY:
The relation between burst and suppression periods in transcranial and direct cortical recorded EEG with cortical amplitudes median nerve somatosensory evoked potentials is studied.

60 patients are included in this study: 15 patients undergoing brain tumor surgery, 15 spine surgery (University Hospital Düsseldorf) and 30 patients during general surgical procedures (Helios Klinikum Wuppertal).

ELIGIBILITY:
Inclusion Criteria:

* Location Helios Klinikum Wuppertal: neurological healthy patients, which undergo an elective surgery under general anaesthesia
* Location Department of Neurosurgery, University Hospital Düsseldorf: all patients with intracranial interventions and the possibility to place a stripe electrode without complications on cortex (it is decided by the surgeon while surgery because of the situs and tumorlocation)

Exclusion Criteria:

* periodical consumption of drugs and pharmaceuticals which influence cortical excitability
* intraoperative contraindication for required depth of anaesthesia
* neurological pre-existing illness
* advanced hepatic insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
SEP ampiltude in burst-suppression-EEG | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Szelényi, Prof., Principal Investigator — Neurosurgical Clinic, Heinrich Heine University
Locations (1):
- Neurosurgical Clinic, Düsseldorf, Germany